CLINICAL TRIAL: NCT06840223
Title: Immediate Effects of Thoracolumbar Fascia Release on Pulmonary Function in Stroke Patients: a Randomized Controlled Study
Brief Title: Thoracolumbar Fascia Release on Pulmonary Function in Stroke
Acronym: TLF-STROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Collaborators: İnönü Üniversitesi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOSTU-25-STROKE-01
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Pulmonary Function; Fascial Manipulation
Keywords: myofascial release; pulmonary function test; spirometry; stroke; thoracolumbar fascia
MeSH Terms: conditions — Stroke | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Traditional stroke rehabilitation (Experimental): Traditional personalized stroke rehabilitation
  Interventions: Other: Traditional stroke rehabilitation
- Thoracolumbar fascia release (Experimental): Traditional personalized stroke rehabilitation plus thorakolumbar fascia release
  Interventions: Other: Thoracolumbar fascia release
- Respiratory exercise (Experimental): Traditional personalized stroke rehabilitation plus respiratory exercise
  Interventions: Other: Respiratory exercise

INTERVENTIONS:
Other: Traditional stroke rehabilitation — Personalized traditional stroke rehabilitation programme including spasticity inhibition, sensory-perceptual-motor integration techniques, core stabilization and strengthening exercises, balance training i.e. applied as needed for stroke patients approximately for 45 minutes
  Arms: Traditional stroke rehabilitation
Other: Thoracolumbar fascia release — Thoracolumbar fascia release was performed by physiotherapist for one session. Supine Pelvic Rotation, Supine Arm Elevation, Bending Forward in Sitting Position and Sitting Crossed Arm and Knee Positions were performed approximately for 10-15 minutes after 45 minutes of traditional stroke rehabilitation.
  Arms: Thoracolumbar fascia release
Other: Respiratory exercise — Respiratory exercises were performed by physiotherapist for one session. Pursed-Lip Breathing, Deep Breathing Exercise, Diaphragm Strengthening Exercise and Thoracic Expansion Exercises were performed approximately for 10-15 minutes after 45 minutes of traditional stroke rehabilitation.
  Arms: Respiratory exercise

SUMMARY:
This study looks at how thoracolumbar fascia release affects breathing in people who had a stroke. After a stroke, many people have trouble breathing well because their muscles become stiff. We want to see if releasing the thoracolumbar fascia (a big sheet of tissue in the lower back) can help improve lung function.

Participants will be divided into three groups:

Control group - Receives standard stroke rehabilitation. Breathing exercise group - Gets standard rehabilitation plus breathing exercises.

Thoracolumbar fascia release group - Gets standard rehabilitation plus thoracolumbar fascia release therapy.

We will measure lung function right after a single session to see if this therapy makes breathing easier.

Our primary outcome is to check if thoracolumbar fascia release improves lung function compared to the other groups.

This study hopes to find new ways to help stroke survivors breathe better and feel more comfortable.

DETAILED DESCRIPTION:
This randomized controlled study investigates the immediate effects of thoracolumbar fascia (TLF) release on pulmonary function in stroke patients. Post-stroke impairments often lead to respiratory dysfunction due to musculoskeletal restrictions and altered neuromuscular control. Given the biomechanical connections between the thoracolumbar fascia and the respiratory system, we hypothesize that TLF release may enhance pulmonary mechanics by improving respiratory functions, in single session.

Participants randomly assigned into three groups:

Control group - Receives standard post-stroke rehabilitation. Respiratory exercise group - Undergoes standard rehabilitation combined with structured breathing exercises.

TLF release group - Receives standard rehabilitation along with thoracolumbar fascia release.

The primary outcome measure is the immediate change in spirometric parameters, including forced vital capacity (FVC%), forced expiratory volume in one second (FEV₁%), FEV₁/FVC (tiffeneu index) and peak expiratory flow (PEF%).

By evaluating the acute effects of thoracolumbar fascial release on respiratory function, this study aims to explore a potential adjunct therapy for post-stroke pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were male patients aged 18-65 years, diagnosed with monohemispheric ischemic stroke above the brainstem, confirmed through computed tomography or magnetic resonance imaging and a stroke diagnosis at least six months prior to the study.

Exclusion Criteria:

Severe cardiorespiratory or neuromuscular disease, tracheostomy, obesity (BMI ≥30 kg/m²), rib cage deformity, cognitive impairment (Mini-Mental State Examination score ≤ 20), and severe dysphagia, aphasia or confusion.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function | From enrollment to the immediately after one session of treatment in all groups
  Spirometric measurements were performed by respiratory physical therapist using COSMED Pony FX spirometer (Elsa Medical Ltd., Rome, Italy) portable device. FEV1(%), FVC (%) and FEV1/FVC and PEF (%) were taken to assess the pulmonary functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Sağlık ve Teknoloji Üniversitesi, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared after ensuring the protection of participants' personal data